CLINICAL TRIAL: NCT05499897
Title: Interscalene Block Relationship With Immunity and Wound Healing
Brief Title: The Effect of Interscalene Block on Wound Healing and Immunity in Open Shoulder Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2022/14
Record Dates: First submitted 2022-08-05; First posted 2022-08-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Ultrasound gıided Interscalene Block
Keywords: peripheral nerve block; general anesthesia; immunity; wound healing
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: This is a randomized,single blind
Who Masked: Participant
Masking Description: Participants will be randomized into 2 groups using the closed envelope method:
  Group GA (Patients who will be operated under general anesthesia): Standard ASA monitoring, induction with 2 mg/kg propofol, 0.6mg/kg rocuronium bromide, 1µcg/kg fentanyl. Maintenance with 2MAC sevoflurane + 40% air mixture. Flow 2L/min. Before extubation, 1 mg/kg tramadol and 15 mg/kg paracetamol will be administered iv. Paracetamol will be repeated at 8 hour intervals.
  Group IS (Patients who will undergo surgery with interscalen block): 20 ml of 0.25% bupivacaine for anesthesia. Before being taken to the postoperative unit, 1 mg/kg tramadol and 15 mg/kg paracetamol will be administered iv. Paracetamol will be repeated at 8 hour intervals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group general anesthesia (Placebo Comparator): (Patients who will be operated under general anesthesia): Standard ASA monitoring, induction with 2 mg/kg propofol, 0.6mg/kg rocuronium bromide, 1µcg/kg fentanyl. Maintenance with 2MAC sevoflurane + 40% air mixture. Flow 2L/min. Before extubation, 1 mg/kg tramadol and 15 mg/kg paracetamol will be administered iv. Paracetamol will be repeated at 8 hour intervals.
  Interventions: Procedure: general anesthesia
- Group interscalene (Experimental): (Patients who will undergo surgery with interscalen block): 20 ml of 0.25% bupivacaine for anesthesia. Before being taken to the postoperative unit, 1 mg/kg tramadol and 15 mg/kg paracetamol will be administered iv. Paracetamol will be repeated at 8 hour intervals.
  Interventions: Procedure: ultrasoud guided interscalene block

INTERVENTIONS:
Procedure: ultrasoud guided interscalene block — Open shoulder surgery by ultrasound guided peripherel block. Observation effect of this peripheral block on immunity and wound healing
  Arms: Group interscalene
Procedure: general anesthesia — Open shoulder surgery by general anesthesia. Observation effect of this peripheral block on immunity and wound healing
  Arms: Group general anesthesia

SUMMARY:
In this study, investigators hypothesize the following: How will the amounts of these factors, which are involved in fibrin formation and wound healing, change after the block? If there is an increase, investigators can conclude that it has a positive effect on wound healing and immunity, if there is no change, it has no effect on wound healing and immunity.

DETAILED DESCRIPTION:
Study design and participants

* 40 participants
* Between 18-65
* ASA physical status I-II
* Scheduled for elective open shoulder surgery
* From July 2022 Exclusion criteria included;
* coagulation disorders
* neuropathic disorders
* diaphragmatic paralysis
* allergy to local anesthetics
* severe cardiopulmonary disease
* psychiatric disorders
* pregnancy
* severe obesity (body mass index >35kg/m2 )
* previous shoulder surgery
* a failed ISB
* liver failure
* kidney failure
* receiving effective treatment on immunity
* Immunosuppression
* Persons requiring intraoperative blood transfusion Randomization

Participants will be randomized into 2 groups using the closed envelope method:

Group GA (Participants who will be operated under general anesthesia): Standard ASA monitoring, induction with 2 mg/kg propofol, 0.6mg/kg rocuronium bromide, 1µcg/kg fentanyl. Maintenance with 2MAC sevoflurane + 40% air mixture. Flow 2L/min. Before extubation, 1 mg/kg tramadol and 15 mg/kg paracetamol will be administered iv. Paracetamol will be repeated at 8 hour intervals.

Group IS (Participants who will undergo surgery with interscalen block): 20 ml of 0.25% bupivacaine for anesthesia. Before being taken to the postoperative unit, 1 mg/kg tramadol and 15 mg/kg paracetamol will be administered iv. Paracetamol will be repeated at 8 hour intervals.

A researcher not associated with the study will apply the random allocation sequence using a computer-generated randomization table. The allocation ratio will be 1:1 and sealed opaque envelopes will be used to conceal the allocations. Outcome assessors, and surgeons will be unaware of the group assignments.

Preoperative Management Before half an hour surgery, blood account will be done for both groups. Platelet count will be done and PDGF (Platelet growth factor), TGF-α (transforming growth factor), EGF (epidermal growth factor), IL-1/IL-2, TNF-α (tumor necrosis factor alpha) will be analysed. The same analyses will be repeated after 24 and 48 hours surgery. These tests will be done 3 times for each patient: preop, postop 24h and postop 48h.

Anesthesia Standard ASA monitors will be used throughout the surgery. Group IS patients will receive a standardized single injection ISB under ultrasound guidance, administered by one of two experienced anesthesiologists (AET or NY). Participants will receive 2mg of midazolam and 50µg of fentanyl for sedation before the block procedure. Each participant will be placed in the supine position with the head turned away from the side to be blocked. A high-frequency linear transducer ultrasound probe will be placed in supraclavicular fossa to identify the subclavian artery and brachial plexus under sterile conditions. 20 ml of 0.25% bupivacaine will be applied with 80mm, 22 gauge needle in-plane technic around the C5 and C6 roots or the superior trunk . Localization will be confirmed by ultrasound visualization of injectate 5mL saline. Before being taken to the postoperative unit, 1 mg/kg tramadol and 15 mg/kg paracetamol will be administered iv. Paracetamol will be repeated at 8 hour intervals.

Group GA participants will be operated under general anesthesia. 2 mg/kg propofol, 0.6mg/kg rocuronium bromide, 1µcg/kg fentanyl will be applied for induction, 2MAC sevoflurane + 40% air mixture for maintenance. Before ekstubation1 mg/kg tramadol iv and 15 mg/kg paracetamol iv will be administered. Paracetamol will be repeated at 8 hour intervals. Participants were extubated in the operating room after reversing residual muscle relaxation.

Postoperative Management All participants will be hospitalized min for 72 hours after surgery. Blood analyses will be done post op 24 and 48 hours. And patients will be called one week later for control. Wound healing will be observed and noted for pain, redness, edema, increased temperature. Findings will be recorded on the follow-up form.

ELIGIBILITY:
Inclusion Criteria:

* 40 patients
* Between 18-65
* ASA physical status I-II
* Scheduled for elective open shoulder surgery

Exclusion Criteria:

* coagulation disorders
* neuropathic disorders
* diaphragmatic paralysis
* allergy to local anesthetics
* severe cardiopulmonary disease
* psychiatric disorders
* pregnancy
* severe obesity (body mass index >35kg/m2 )
* previous shoulder surgery
* a failed ISB
* liver failure
* kidney failure
* receiving effective treatment on immunity
* Immunosuppression
* Persons requiring intraoperative blood transfusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 40 patients, Between 18-65, males and females
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
interscalene block | 6 monthes
  number of participants with interscalene block

SECONDARY OUTCOMES:
general anesthesia | 6 monthes
  Number of participants with general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Arzu E Tekeli, MD, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van Yüzüncü Yil University, Van, Bardakçı, Turkey (Türkiye)